CLINICAL TRIAL: NCT01920984
Title: Vitreous Levels of Cysteine-rich 61 in Patients With Proliferative Diabetic Retinopathy
Acronym: VL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: NSC96-2628-B-002-032-MY3
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2004-01

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pretreatment of bevacizumab (Experimental): Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) 7 to 9 days before vitrectomy due to diabetic retinopathy.
  Interventions: Drug: intravitreal injection of 1.25 mg of bevacizumab
- No pretreatment of bevacizumab (No Intervention): Patients will not receive bevacizumab pretreatment before vitreous surgery.

INTERVENTIONS:
Drug: intravitreal injection of 1.25 mg of bevacizumab — Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) 7 to 9 days before vitrectomy
  Other Names: Bevacizumab(Avastin, Genentech, Inc., South San Francisco)
  Arms: pretreatment of bevacizumab

SUMMARY:
To determine the vitreous levels of fractalkine, cysteine-rich 61 (Cyr61), and VEGF in patients with PDR. Verifying that it is greater to that found in non-diabetic patients with different non-angiogenetic diseases.

DETAILED DESCRIPTION:
Introduction:

Angiogenesis, the growth and proliferation of new blood vessels, is an important aspect of the vascular proliferation found in tumor growth, wound repair, inflammatory states, and ischemic sequel in the ocular angiogenetic diseases. Intraocular neovascularization, the major eventually complication of diabetic mellitus, may result in vitreous hemorrhage, tractional retinal detachment, neovascularization glaucoma and eventually blindness. The involved factors include basic fibroblast growth factor (bFGF), insulin-like growth factor-I (IGF-I), vascular endothelial cell growth factor (VEGF), and Connective tissue growth factor (CTGF)/Cysteine-rich protein (Cyr61)/Nephroblastoma overexpressed gene (CCN) family. VEGF is a primary angiogenic factor that mediates ischemic-induced retinal neovascularization. VEGF level are elevated in the vitreous fluid in patients with proliferative diabetic retinopathy (PDR). The unselective anti-VEGF antibody bevacizumab has been used for the treatment of diabetic retinopathy.

Problem:

In spite of its potent anti-VEGF property, it does not completely inhibit ischemia-induced retinal neovascularization. Several other factors which were detected to have increased vitreous levels in the PDR patients might participate in the angiogenic process of diabetic retinopathy. One of the member of the CCN family, connective tissue growth factor (CTGF), was found to be involved in the angiogenesis and fibrosis mechanism of PDR. It is unclear if the other factors in the CCN family might also control the development of retinal angiogenesis and fibrosis.We measured vitreous cysteine-rich 61 (Cyr61) levels in PDR patients, non-diabetic patients,and PDR patients pretreated with bevacizumab. We further correlated the cysteine-rich 61 levels with different stages of PDR. Concomitant VEGF level was also measured to better understand the interaction of different factors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with type 1 or type 2 diabetes mellitus
* Not eligible for any currently approved treatments or experimental protocols
* Patients with PDR who receiving vitreoretinal surgery.

Exclusion Criteria:

* A condition that would preclude a patient for participation in the study in opinion of investigator, e.g., unstable medical status including glycemic control and blood pressure
* Panretinal laser photocoagulation in the study eye
* Previous treatment with intravitreal or sub-Tenon triamcinolone
* History of submacular surgery or other surgical intervention for diabetic

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Vitreous levels of Fractalkine, Cyr61, and VEGF of patients with proliferative diabetic retinopathy | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hao Yang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Watanabe D, Suzuma K, Matsui S, Kurimoto M, Kiryu J, Kita M, Suzuma I, Ohashi H, Ojima T, Murakami T, Kobayashi T, Masuda S, Nagao M, Yoshimura N, Takagi H. Erythropoietin as a retinal angiogenic factor in proliferative diabetic retinopathy. N Engl J Med. 2005 Aug 25;353(8):782-92. doi: 10.1056/NEJMoa041773. PMID 16120858